CLINICAL TRIAL: NCT05294874
Title: Gait Rehabilitation in Ambulant Diplegic Children Using BOTOX and Ankle Weights
Brief Title: Gait Rehabilitation in Diplegic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ibrahim, lecturer physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pediatrics
Record Dates: First submitted 2022-03-06; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy; Spastic Diplegia
Keywords: gait; diplegia; ankle weight; botox injection
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- classical gait training (Active Comparator): physical therapy exercises including classical gait training
  Interventions: Other: gait training
- classical gait training using ankle weight (Active Comparator): physical therapy exercises including classical gait training while using ankle weight
  Interventions: Other: gait training
- gait training using ankle weight after botulinum toxin injection (Experimental): physical therapy exercises including classical gait training while using ankle weight and with BOTOX injection
  Interventions: Other: gait training

INTERVENTIONS:
Other: gait training — walking forward, sideway and backward walking on balance board
  Other Names: rehabilitation

SUMMARY:
Background: Standing and walking serve an individual's basic need to move from place to place, and both are the most common activities that people do on a daily basis.

Aim: to investigate the combined effect of botulinum toxin A (BoNT-A) injection and ankle weight on the gait of diplegic children who are using Ankle foot orthoses.

DETAILED DESCRIPTION:
Methods: Sixty children with spastic diplegia were included in this prospective, controlled trial. Children were divided into three groups, each with 20 patients: Group 1 received classical gait rehabilitation; Group 2 received the same gait training while adding ankle weight ; and Group 3 received the same as group 2 plus botulinum toxin injection. The Modified Ashworth Scale (MAS),knee range-of-motion measures, and Hoffman /Myogenic reflex ratio were used to examine patients before the commencement of treatment and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as spastic diplegia.
* They were able to follow simple verbal instructions.
* The use of Ankle Foot Orthoses.
* Spasticity grade of 1+ or 2 in both calf and hamstring muscles according to modified Ashworth's scale (MAS).
* level I or II on the Gross Motor Function Classification System (GMFCS).

Exclusion Criteria:

* fixed contractures or deformities in the lower limbs.
* surgical orthopedic intervention.
* Botulinum A injection or use of neuromuscular blockers in the previous 6 months before the start of study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
measurement of knee excursion during gait | after 3 months of the treatment program.
  evaluation of knee flexion range of motion during gait using two dimension gait analysis.
evaluation of spasticity: modified ashowrth scale scores | after 3 months of the treatment program.
  hamstring and calf muscles evaluation of spasticity through passive movement .the score ranged from 0 ( nearly normal) to 5 (rigid in flexion or extension)

SECONDARY OUTCOMES:
electromyography to asses spasticity in hamstring and calf muscles | after 3 months of the treatment program.
  Hoffman/Myogenic reflex to assess spasticity ratio

CONTACTS AND LOCATIONS:
Overall Officials: Nahla mohamed, phd, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy,Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
tables and figures of statistical analysis published
Supporting Information: Study Protocol, SAP
Time Frame: after publication of the results
Access Criteria: through contact the authors